CLINICAL TRIAL: NCT01359124
Title: Reaching Exercise Goals: Comparison of the Underwater Treadmill, Land Based Treadmill, and Exercise Cycle in Patients With Knee Osteoarthritis
Brief Title: Reaching Exercise Goals: Comparison of Exercise Means in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, April Armstrong, Associate Professor, Milton S. Hershey Medical Center
Other Study IDs: IRB#35938
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Exercise Therapies
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Plyometric Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Water Treadmill: These subjects will participate in three monitored exercise sessions per week for 8 weeks using a water-based treadmill.
  Interventions: Behavioral: Water-based Treadmill
- Land Treadmill: These subjects will participate in three monitored exercise sessions per week for 8 weeks using a land-based treadmill.
  Interventions: Behavioral: Land-based Treadmill
- Exercise Cycle: These subjects will participate in three monitored exercise sessions per week for 8 weeks using an upright exercise cycle.
  Interventions: Behavioral: Exercise Cycle

INTERVENTIONS:
Behavioral: Exercise Cycle — Exercise regimen: three monitored exercise sessions per week for eight weeks using the upright exercise cycle.
  Other Names: Schwinn Windsprint Exercise Cycle
  Groups: Exercise Cycle
Behavioral: Land-based Treadmill — Exercise regimen: three monitored exercise sessions per week for eight weeks using the land-based treadmill.
  Other Names: True CS 6.0 treadmill; Nautilus NTR 700 treadmill
  Groups: Land Treadmill
Behavioral: Water-based Treadmill — Exercise regimen: three monitored exercise sessions per week for eight weeks using the water-based treadmill.
  Other Names: Hydroworx 2000 Series pool treadmill
  Groups: Water Treadmill

SUMMARY:
The primary objective is to evaluate water based treadmill exercise, land based treadmill exercise, and upright cycling in meeting American College of Sports Medicine exercise goals for moderate exercise.

The secondary objective is to compare exercise tolerance for water based treadmill, land based treadmill, and upright cycling in meeting American College of Sports Medicine exercise goals for moderate exercise.

The tertiary objective is to evaluate quality of life improvements for water based treadmill exercise, land based treadmill exercise, and upright cycling.

DETAILED DESCRIPTION:
Osteoarthritis is the most common joint disorder in the United States, affecting approximately 26.9 million adults greater than 25 years of age. This disorder can be very debilitating: more than 40% of adults with doctor diagnosed arthritis have reported that joint symptoms cause them to modify their activities. Risk of disability (defined as needing help walking or climbing stairs) associated with osteoarthritis is considered equivalent to cardiovascular disease and is greater than any other medical condition in elderly patients [13]. Persons with disability associated with osteoarthritis have a substantially worse health-related quality of life, in large part due to their inability to exercise.

Exercise has been shown to help maintain function in knee osteoarthritis [5]. Aerobic walking and quadriceps strengthening exercises ([18];[7]) and resistance training [15] have demonstrated that exercise can potentially improve pain and function in individuals with knee osteoarthritis. Likewise, a Cochrane review on aquatic exercise provided gold level evidence that aquatic exercise probably reduces pain and increases function over 3 months; but, it stated clearly that more research was needed to understand which type of aquatic exercise, how often, and for how long might be beneficial [2]. The American College of Sports Medicine (ACSM) recommendations for healthy adults recommend moderate-intensity aerobic exercise (endurance) physical activity for a minimum of 30 minutes, 5 days per week or vigorous-intensity aerobic physical activity for a minimum of 20 minutes, 3 days per week in all healthy adults aged 18 to 65 to promote and maintain health [9]. The best method of reaching current ACSM goals in patients with knee osteoarthritis is not known, as impact-related exercise certainly demands healthy joints and many patients with knee osteoarthritis do not tolerate this form of exercise.

In counseling patients with knee osteoarthritis, the question remains: how best to exercise to reach the ACSM goals for exercise. This study will compare water-based and land-based treadmill exercise and upright cycling in meeting ACSM exercise goals for moderate exercise.

Interested subjects will undergo knee radiographs to confirm presence and degree of knee osteoarthritis. Eligible participants will then be randomized into one of the three exercise cohorts. During each session, participants will complete between 10 to 45 minutes of exercise, with a goal of achieving 30 minutes of moderate aerobic exercise. All subjects will only participate in routine activities for the 8 week study period outside of the study protocol (no strength training, cardio training, etc.). Health status measurement questionnaires (WOMAC, KOOS, and SF12) will be completed at the time of randomization and at the conclusion of each week of exercise for a total of 9 times.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30-60
* Knee pain
* Radiographically confirmed knee osteoarthritis

Exclusion Criteria:

* Medical conditions contraindicating moderate aerobic exercise as determined through prescreening questions, ie: heart condition, asthma, history of stroke.
* Inability to exercise via treadmill or exercise cycle
* Contraindication to radiography
* Pregnancy
* History of recent joint injection (steroid, synvisc, etc.) within 6 weeks of study
* History of previous joint arthroplasty
* History of inflammatory joint disease
* Inability to sign informed consent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects for this study will be recruited from Penn State Milton S. Hershey Medical Center and surrounding communities via internal and external advertisements.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Exercise Tolerance | 8 weeks
  Exercise tolerance will be assessed based upon changes in symptoms related to knee osteoarthritis and exercise limitations related to those symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Silvis, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Ainsworth BE, Haskell WL, Whitt MC, Irwin ML, Swartz AM, Strath SJ, O'Brien WL, Bassett DR Jr, Schmitz KH, Emplaincourt PO, Jacobs DR Jr, Leon AS. Compendium of physical activities: an update of activity codes and MET intensities. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S498-504. doi: 10.1097/00005768-200009001-00009. PMID 10993420
- [Background] Bartels EM, Lund H, Hagen KB, Dagfinrud H, Christensen R, Danneskiold-Samsoe B. Aquatic exercise for the treatment of knee and hip osteoarthritis. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD005523. doi: 10.1002/14651858.CD005523.pub2. PMID 17943863
- [Background] Bosomworth NJ. Exercise and knee osteoarthritis: benefit or hazard? Can Fam Physician. 2009 Sep;55(9):871-8. PMID 19752252
- [Background] Cottrell E, Roddy E, Foster NE. The attitudes, beliefs and behaviours of GPs regarding exercise for chronic knee pain: a systematic review. BMC Fam Pract. 2010 Jan 18;11:4. doi: 10.1186/1471-2296-11-4. PMID 20082694
- [Background] Dunlop DD, Semanik P, Song J, Sharma L, Nevitt M, Jackson R, Mysiw J, Chang RW; Osteoarthritis Initiative Investigators. Moving to maintain function in knee osteoarthritis: evidence from the osteoarthritis initiative. Arch Phys Med Rehabil. 2010 May;91(5):714-21. doi: 10.1016/j.apmr.2010.01.015. PMID 20434608
- [Background] Dunn AL, Jewell JS. The effect of exercise on mental health. Curr Sports Med Rep. 2010 Jul-Aug;9(4):202-7. doi: 10.1249/JSR.0b013e3181e7d9af. PMID 20622537
- [Background] Ettinger WH Jr, Burns R, Messier SP, Applegate W, Rejeski WJ, Morgan T, Shumaker S, Berry MJ, O'Toole M, Monu J, Craven T. A randomized trial comparing aerobic exercise and resistance exercise with a health education program in older adults with knee osteoarthritis. The Fitness Arthritis and Seniors Trial (FAST). JAMA. 1997 Jan 1;277(1):25-31. PMID 8980206
- [Background] Fransen M, McConnell S. Exercise for osteoarthritis of the knee. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD004376. doi: 10.1002/14651858.CD004376.pub2. PMID 18843657
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Heckman GA, McKelvie RS. Cardiovascular aging and exercise in healthy older adults. Clin J Sport Med. 2008 Nov;18(6):479-85. doi: 10.1097/JSM.0b013e3181865f03. PMID 19001881
- [Background] Helmick CG, Felson DT, Lawrence RC, Gabriel S, Hirsch R, Kwoh CK, Liang MH, Kremers HM, Mayes MD, Merkel PA, Pillemer SR, Reveille JD, Stone JH; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part I. Arthritis Rheum. 2008 Jan;58(1):15-25. doi: 10.1002/art.23177. PMID 18163481
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Hunter DJ, McDougall JJ, Keefe FJ. The symptoms of osteoarthritis and the genesis of pain. Rheum Dis Clin North Am. 2008 Aug;34(3):623-43. doi: 10.1016/j.rdc.2008.05.004. PMID 18687276
- [Background] Kotlarz H, Gunnarsson CL, Fang H, Rizzo JA. Insurer and out-of-pocket costs of osteoarthritis in the US: evidence from national survey data. Arthritis Rheum. 2009 Dec;60(12):3546-53. doi: 10.1002/art.24984. PMID 19950287
- [Background] Lange AK, Vanwanseele B, Fiatarone Singh MA. Strength training for treatment of osteoarthritis of the knee: a systematic review. Arthritis Rheum. 2008 Oct 15;59(10):1488-94. doi: 10.1002/art.24118. PMID 18821647
- [Background] Lee IM. Physical activity and cardiac protection. Curr Sports Med Rep. 2010 Jul-Aug;9(4):214-9. doi: 10.1249/JSR.0b013e3181e7daf1. PMID 20622539
- [Background] Roddy E, Zhang W, Doherty M. Aerobic walking or strengthening exercise for osteoarthritis of the knee? A systematic review. Ann Rheum Dis. 2005 Apr;64(4):544-8. doi: 10.1136/ard.2004.028746. PMID 15769914
- [Background] Schiphof D, Boers M, Bierma-Zeinstra SM. Differences in descriptions of Kellgren and Lawrence grades of knee osteoarthritis. Ann Rheum Dis. 2008 Jul;67(7):1034-6. doi: 10.1136/ard.2007.079020. Epub 2008 Jan 15. PMID 18198197
- [Background] Whaley MH, Brubaker PH, Otto RM. ACSM's Guidelines for Exercise Testing and Prescription, 7th edition. USA: Lippincott Williams and Wilkins, 2006, pgs. 77-78, 146.
- [Background] Wyatt FB, Milam S, Manske RC, Deere R. The effects of aquatic and traditional exercise programs on persons with knee osteoarthritis. J Strength Cond Res. 2001 Aug;15(3):337-40. PMID 11710661
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Rheum Dis Clin North Am. 2008 Aug;34(3):515-29. doi: 10.1016/j.rdc.2008.05.007. PMID 18687270